CLINICAL TRIAL: NCT07001800
Title: A Phase 2b/3, Randomized, Double-Blinded, Placebo Controlled Study ChecKing the Efficacy and Safety of ATAciguat to Slow the Progression of VaLvular DYsfunction in Participants With Moderate Calcific Aortic Valve STenosis
Brief Title: Ataciguat for Slowing the Progression of Moderate Calcific Aortic Valve Stenosis: A Randomized, Placebo Controlled Study
Acronym: KATALYST-AV
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kardigan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATA-301
Record Dates: First submitted 2025-05-13; First posted 2025-06-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Moderate Aortic Valve Stenosis
Keywords: Ataciguat; sGC activator; sGC stimulator; Aortic valve stenosis; Moderate aortic valve stenosis; Calcific aortic valve stenosis; CAVS; Moderate Calcific Aortic Valve Stenosis; Aortic Stenosis (AS)
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — 5-chloro-2-(5-chlorothiophene-2-sulfonylamino)-N-(4-(morpholine-4-sulfonyl)phenyl)benzamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ataciguat (Experimental)
  Interventions: Drug: Ataciguat
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ataciguat — Ataciguat will be administrated daily for up to 156 weeks
  Arms: Ataciguat
Drug: Placebo — Placebo will be administrated daily for up to 156 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate if ataciguat slows the progression of moderate calcific aortic valve stenosis in adults.

DETAILED DESCRIPTION:
This study will be conducted in two parts: Part A and Part B. The purpose of Part A is to investigate whether ataciguat slows the progression of aortic valve calcium (AVC) deposition in adults with moderate calcific aortic valve stenosis (CAVS). The safety, tolerability, and pharmacokinetics of ataciguat will also be evaluated. Approximately 132 participants will be enrolled in Part A. Enrollment in Part B will begin once enrollment in Part A is complete. The purpose of Part B is to investigate whether ataciguat slows the rate of aortic valve area (AVA) loss and to evaluate the effect of ataciguat on peak oxygen consumption (VO2) in participants with moderate CAVS. The safety and tolerability of ataciguat will also be evaluated. Approximately 1144 participants will be enrolled in Part B.

ELIGIBILITY:
Key Inclusion Criteria:

1. Adult male or female at least 50 years of age
2. Has moderate CAVS as defined by:

   1. An AVA of ≥1.0 cm2 to ≤1.50 cm2
   2. An AVC score between ≥600 to 1200 Agatston units (AU) for women and between ≥600 to 2000 AU for men
3. Has a left ventricular ejection fraction (EF) of ≥45% at the time of Screening as determined by the echocardiography Imaging Core Laboratory
4. For participants on beta blockade, the dose must be stable for at least 90 days prior to the Screening Visit with no anticipated changes during the study

Key Exclusion Criteria:

1. For participants in the CPET sub-study in Part A and all participants in Part B: Has any medical or physical condition that, in the Investigator's opinion, could lead to an inability to complete Protocol-required CPET procedures (eg, pulmonary disease, joint, leg, hip, back conditions that limit physical activity, or other absolute contraindications for CPET)
2. Anticipated or planned prior aortic valve replacement, repair, surgery, or intervention in the next 6 months
3. Has moderate, moderate-to-severe, or severe (Grade 2 or higher) mitral stenosis, mitral regurgitation, and/or aortic regurgitation
4. Has suspected or known congenital aortic valve disease including bicuspid aortic valve
5. New York Heart Association (NYHA) Class III or Class IV
6. Has a primary etiology for heart failure other than aortic valve disease
7. Has coronary artery disease or anticipating coronary stenting surgery
8. Abnormal electrocardiogram (ECG) results or long-standing persistent or permanent atrial fibrillation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1276 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
(Part A) Change in Aortic Valve Calcium (AVC) score as assessed by non-contrast CT from baseline to Week 24 | Week 24
(Part B Dual-Primary) Percent change in Aortic Valve Area (AVA) as measured by echocardiogram from baseline to Week 48 | Week 48
(Part B Dual-Primary) Change in peak VO2 by CPET from baseline to Week 48 | Week 48

SECONDARY OUTCOMES:
(Part A) Correlation in the change in AVC as assessed by non-contract CT and change in VO2 as assessed be remote cardiac monitoring devices at Week 48 | Week 48
(Part A) Change in VO2 as assessed by remote cardiac monitoring devices from baseline to Week 48 | Week 48
(Part A) Change in Left Ventricular Mass Index (LVMI) from baseline to Week 48 | Week 48
(Part A) Change in Kansas City Cardiomyopathy Questionnaire-23 (KCCQ-23) from baseline to Week 48 | Week 48
  KCCQ-23 is a patient reported outcome instrument with minimum score = 0 and maximum score = 100 where higher score indicates better health status. There are no units to the score.
(Part B) Change in AVC score as assessed by non-contrast CT from baseline to Week 48 | Week 48
(Part B) Time to decision to proceed with TAVR/SAVR or all-cause death | Week 158
(Part B) Percentage of participants with progression to AVA <1.0cm2 at Week 48 | Week 48

CONTACTS AND LOCATIONS:
Locations (58):
- United States (58):
  - University of Alabama at Birmingham (UAB) - Medical Center, Birmingham, Alabama
  - Heart Center Research LLC, Huntsville, Alabama
  - Onyx Clinical Research - Peoria, Peoria, Arizona
  - National Heart Institute, Beverly Hills, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Profound Research LLC at Southern California Heart Specialists, Pasadena, California
  - University of California, San Francisco (UCSF) - Medical Center, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor UCLA Medical Center, Torrance, California
  - HCA Florida - JFK Hospital, Atlantis, Florida
  - New Generation of Medical Research, Hialeah, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - New Generation of Medical Research - Naples, Naples, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Northwestern University The Feinberg School of Medicine, Chicago, Illinois
  - NorthShore University Health System, Glenview, Illinois
  - Midwest Cardiovascular Institute, Naperville, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - St. Vincent Medical Group, Inc., Carmel, Indiana
  - University of Iowa Health Care, Iowa City, Iowa
  - University of Louisville Health, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Corewell Health, Royal Oak, Michigan
  - Henry Ford Hospital, West Bloomfield, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Atlantic Health System - Morristown Medical Center, Morristown, New Jersey
  - Inspira Medical Center of Vineland, Vineland, New Jersey
  - Albany Medical Center, Albany, New York
  - University of Buffalo, Buffalo, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University School of Medicine, Durham, North Carolina
  - Moses H. Cone Memorial Hospital Operating Corporation d/b/a Cone Health, Greensboro, North Carolina
  - Sanford Fargo, Fargo, North Dakota
  - The Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ascension St. John Jane Phillips Hospital, Bartlesville, Oklahoma
  - Ascension St. John Hospital, Tulsa, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - OnSite Clinical Solutions, LLC - Rock Hill, Rock Hill, South Carolina
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - Ascension Saint Thomas Heart Midtown, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - St. David's Heart and Vascular dba Austin Heart - Main Office, Austin, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Baylor Scott and White - The Heart Hospital Baylor Plano, Plano, Texas
  - Methodist Hospital - San Antonio, San Antonio, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - University of Utah Hospital & Clinics, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No